CLINICAL TRIAL: NCT04689230
Title: Comparison of the Efficacy Between Small Incision Technique and Upper Blepharoplasty in Treatment of Upper Eyelid Medial Pad Fat Bulge
Brief Title: Small Incision Technique Versus Upper Blepharoplasty in Upper Eyelid Medial Pad Fat Removal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tarek Roshdy mohamed Mahgoub ELhamaky, Lecturer, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hamaky 8
Record Dates: First submitted 2020-12-28; First posted 2020-12-30 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Eyelid Diseases
Keywords: upper eyelid pad fat; blepharoplasty
MeSH Terms: conditions — Eyelid Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- upper eyelid blepharoplasty (Active Comparator): traditional upper eyelid blepharoplasty : upper eyelid entire length incision followed by proper dissection medially to medial pad fat.
  medial pad fat identification and excision. closure of the wound with subcuticular 6/0 vicryl suture
  Interventions: Procedure: upper eyelid blepharoplasty
- small incision technique (Experimental): medial upper eyelid 4 mm length incision followed by proper dissection medially to medial pad fat.
  medial pad fat identification and excision. closure of the wound with interrupted 6/0 vicryl sutures
  Interventions: Procedure: upper eyelid blepharoplasty

INTERVENTIONS:
Procedure: upper eyelid blepharoplasty — upper eyelid blepharoplasty

SUMMARY:
Medial upper eyelid pad of fat bulge is a common problem. Small incision surgery could be a time-efficient, minimally invasive and scar formation procedure .

DETAILED DESCRIPTION:
Traditional upper eyelid blepharoplasty: an entire length upper eyelid crease followed by proper dissection are applied . identification and removal of medial pad of fat.

Small Incision technique: 4 mm medial upper eyelid small incision followed by proper dissection to gain direct access to the medial fat pad removal

ELIGIBILITY:
Inclusion Criteria:

* upper eyelid medial pad of fat bulge

Exclusion Criteria:

Other eyelid diseases and previous eyelid surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-11-15 (Estimated)

PRIMARY OUTCOMES:
global aesthetic improvement scale | 3 months
  calculate scale score (1-5);score 1:exceptional improvement and score 5 :worsened patient

SECONDARY OUTCOMES:
duration of surgery | 3 months
  time of surgery in minutes measured by stopwatch

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Elahamky, M.D., Principal Investigator — Benha university faculty of medicine
Locations (1):
- INMC, Abu Dhabi, United Arab Emirates